CLINICAL TRIAL: NCT05228743
Title: A Randomized, Multicenter, Controlled Study to Compare Hyperthermic Intraperitoneal Chemotherapy Plus Paclitaxel IP/IV, S-1 and Paclitaxel IP/IV，S-1 as Conversion Therapy for Gastric Cancer Patients With Peritoneal Metastasis
Brief Title: Conversion Therapy of Hyperthermic Intraperitoneal Chemotherapy Plus Chemotherapy and Chemotherapy in Stage IV Gastric Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E20201130
Record Dates: First submitted 2020-11-30; First posted 2022-02-08 (Actual); Last update posted 2022-02-08 (Actual); Status verified 2021-09

CONDITIONS: Gastric Cancer
Keywords: conversion therapy; HIPEC; peritoneal metastasis
MeSH Terms: conditions — Stomach Neoplasms | interventions — Hyperthermic Intraperitoneal Chemotherapy; Paclitaxel; S 1 (combination)

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HIPEC plus Paclitaxel IP/IV, S-1 (Experimental): After laparoscopic exploration, HIPEC was started immediately, at least 4 HIPEC was completed.Three to six weeks after HIPEC was completed, chemotherapy was started.The curative effect was evaluated every 2-4 cycles. If the operation standard of R0 was met, the second laparoscopic staging was performed: if the peritoneal metastasis reached P 0 or P1a, the operator judged that R0 could be removed. Open radical gastrectomy (D2 / D2 +) was performed. For P1b / c cases, the original treatment was continued until the disease progressed.
  Interventions: Procedure: Comparing Hyperthermic Intraperitoneal Chemotherapy; Drug: Paclitaxel; Drug: S1
- Paclitaxel IP/IV, S-1 (No Intervention): Within one week after laparoscopic exploration, chemotherapy was started. The curative effect was evaluated every 2-4 cycles. If the operation standard of R0 was met, the second laparoscopic staging was performed: if the peritoneal metastasis reached P 0 or P1a, the operator judged that R0 could be removed. Open radical gastrectomy (D2 / D2 +) was performed. For P1b / c cases, the original treatment was continued until the disease progressed.

INTERVENTIONS:
Procedure: Comparing Hyperthermic Intraperitoneal Chemotherapy — After laparoscopic exploration, HIPEC was started immediately: the temperature was 43 ℃ and the duration was 60 min. paclitaxel (PTX) was used with a dose of 50mg / m2. The second HIPEC was completed 24-48 hrs after the first HIPEC, and at least 4 HIPEC was completed.
  Other Names: HIPEC
  Arms: HIPEC plus Paclitaxel IP/IV, S-1
Drug: Paclitaxel — A natural anticancer drug that has been widely used in the treatment of breast, ovarian and some head and neck and lung cancers.Three to six weeks after HIPEC was completed, chemotherapy was started:: PTX: 50mg / m2 IV, D1, D8; PTX: 20mg / m2 IP, D1, D8; q3w; S-1: 60mg / m2, bid, d1-14, repeated every 3 weeks.
  Other Names: PTX
  Arms: HIPEC plus Paclitaxel IP/IV, S-1
Drug: S1 — S-1 is an oral fluoropyrimidine consisting of tegafur (a prodrug that is converted to fluorouracil, mainly in liver microsomes but also in tumour tissue), gimeracil (an inhibitor of dihydropyrimidine dehydrogenase, which degrades 5-FU), and oteracil (which inhibits the phosphorylation of 5-FU in the gastrointestinal tract, thereby reducing the toxic effects of 5-FU in the intestinum).Three to six weeks after HIPEC was completed, chemotherapy was started:: PTX: 50mg / m2 IV, D1, D8; PTX: 20mg / m2 IP, D1, D8; q3w; S-1: 60mg / m2, bid, d1-14, repeated every 3 weeks.
  Arms: HIPEC plus Paclitaxel IP/IV, S-1

SUMMARY:
The main purpose of this study is to compare Hyperthermic Intraperitoneal Chemotherapy combined with Chemotherapy and Chemotherapy as a conversion therapy for gastric Cancer Patients with peritoneal metastasis in Safety and Effectiveness.

DETAILED DESCRIPTION:
Follow-up results from the PHOENIX study failed to show statistical superiority of intraperitoneal paclitaxel plus systemic chemotherapy. However, in the subgroup analysis, it can be seen that after correcting for the bias effect of ascites, the difference between the two groups was statistically significant, further proving the significance of ascites control on the prognosis of patients with gastric cancer peritoneal metastasis. Based on the existing data, for patients with moderate amount of ascites, the IP regimen is recommended to control ascites and relieve ascites. Symptoms, purpose of improving quality of life and prolonging survival. HIPEC is traditionally used to treat peritoneal cancer. Patients who diagnosed with gastric cancer with peritoneal metastasis were divided into two groups based on whether they underwent HIPEC. The primary endpoint is the R0 resection rate and the secondary endpoints are 1-year overall survival, and Safety.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed as gastric adenocarcinoma by pathology and had not received any other anti-tumor treatment such as radiotherapy and chemotherapy;
* ≥ 18 and ≤ 70 years of age; Eastern Cooperative Oncology Group Performance Status (ECOG): 0-1;
* Intraoperative pathological diagnosis was peritoneal metastasis (stage ≤ P1b), with or without ascites (ascites volume exceeding pelvic cavity but not reaching full abdominal ascites)
* Patients have adequate baseline organ and marrow function :hemoglobin≥9g/dL; absolute neutrophil count (ANC) ≥1,500/mm3; PLT(platelets)≥1000,000/mm3; total bilirubin ≤1.5×upper normal limit(ULN); AST ≤2.5 ×ULN, ALT ≤2.5 ×ULN; prothrombin time-international normalized ratio≤1.5, and APTT(activated partial thromboplastin time) was within normal range; creatine ≤ 1.5 x ULN;
* Written informed consent provided;

Exclusion Criteria:

* Diagnosed as Her-2(+++)/FISH(+) by pathology;
* With other distant metastasis(ovarian metastasis was excluded)
* Patients with Serious liver disease (such as cirrhosis, etc.), kidney disease, respiratory disease or uncontrolled diabetes, hypertension and other chronic systemic diseases, heart disease with Clinical symptoms, such as congestive heart failure, coronary heart disease symptoms, drug is difficult to control arrhythmia, hypertension, or six months had a myocardial infarction attack, or cardiac insufficiency;
* Organ transplantation patients need immunosuppressive therapy;
* Severe recurrent infections were not controlled or with other serious concomitant diseases;
* Patients got other primary malignant tumors (except curable skin basal cell carcinoma and cervical cancer in situ) except gastric cancer within 5 years; Psychiatric disease which require treatment;
* Within 6 months before study starts and in the process of this study, patients participate in other clinical researches;
* Patients with peripheral nervous system disorder or apparent mental disorders or had the history of central nervous system disorders;
* Pregnant or lactating women, women of child-bearing potential, unwilling to use adequate contraceptive protection during the process of the study;
* Patients without legal capacity,or medical/ethical reasons may influence the study to continue.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2023-08-31 (Estimated); Study Completion 2023-10-31 (Estimated)

PRIMARY OUTCOMES:
R0 resection rate | 1 year

SECONDARY OUTCOMES:
1 year overall survival | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Gastrointestinal Medical Oncology, Tianjin Medical University Cancer Hospital, Tianjin, Tianjin Municipality, China